CLINICAL TRIAL: NCT02855723
Title: Randomized, Open-label Economic and Medical Study on the Lymph Node Management of Squamous Cell Carcinoma of the Oral Cavity and Oropharynx T1-T2N0 Operable : Comparison of the Reference Strategy Based on a the Systematic Lymph Node Dissection Versus the Strategy Based on the Technique of Sentinel Lymph Node.
Brief Title: Randomized, Open-label Economic and Medical Study on the Lymph Node Management of Squamous Cell Carcinoma of the Oral Cavity and Oropharynx Tumor Stage 1 or 2, Nodes 0 (T1-T2 N0) Operable
Acronym: SentiMERORL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF 5023; 2007- AO1191-52 (Other: Afssaps - Agence française de sécurité sanitaire des produits de santé (Saint-Denis))
Record Dates: First submitted 2016-07-19; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Head and Neck Tumors
Keywords: Squamous carcinoma of oral cavity and oropharynx; Sentinel lymph node; Lymph node dissection; Equivalence
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GS strategy (Active Comparator): sentinel node biopsy
  Interventions: Other: Surgery: GS strategy
- Classic strategy (Other): systematic lymphadenectomy
  Interventions: Other: Surgery: Classic strategy

INTERVENTIONS:
Other: Surgery: GS strategy — sentinel node biopsy
  Arms: GS strategy
Other: Surgery: Classic strategy — systematic lymphadenectomy
  Arms: Classic strategy

SUMMARY:
Currently, patients with cancer of oral cavity or oropharynx T1-T2N0 classified, are treated surgically with systematic lymph node dissection while in 70%, there is no lymph node metastasis. The technique of identifying the sentinel node (GS) is validated for these tumors because the status of the sentinel node is predictive of the other nodes status in the neck. This helps to diagnose the presence of metastases without lymph node dissection and thus select patients requiring a treatment node. However, the oncological and functional results of a therapeutic strategy based on identifying the GS is unknown.

This open-label randomized multicenter clinical trial aims to compare the oncologic and functional outcome of two strategies : the current management versus the management based on the sentinel lymph node.

The hypothesis is based on a nodal control difference at 2 years in both arms not exceeding 10%. The medico-economic analysis will be conducted in two stages : a classic stage on 2 years with estimated incremental cost-effectiveness and incremental cost-utility, then a step with log term modeling.

A reduction in morbidity and treatment costs in the sentinel node arm are expected in this study.

DETAILED DESCRIPTION:
This study schedules the screening visit (V0) and then 9 follow-up visits during 24 months.

At the screening, after verification of the eligibility criteria and signature of the informed consent form, the subject will be randomized in one of 2 arms. At the inclusion the following exams have to be done : clinical exam, panendoscopy, cytologic and histologic analysis and CT-Scan (or MRI). For each visit, the investigator will perform a clinical exam and the subjects should complete some questionnaires themselves from V0 to V3, V6 (12 months) and V9. At the last visit (24 months) the patients will have a CTC-Scan ou MRI.

At the end of the follow-up period (24 months), the data of subjects survival will be recorded during three years.

ELIGIBILITY:
Inclusion criteria:

1. Man or woman age over 18 without upper age limit
2. Social Insured
3. Patient Information and Informed Consent signed by the patient
4. Patient not participating in another trial since the legal time
5. Absence of any previous treatment for cancer of the Upper AeroDigestive Tract (VADS)
6. Patient with primary squamous cell carcinoma of the oral cavity or oropharynx documented by biopsy with histopathologic analysis not older than 1 month
7. curable or operable tumor with radiation under the Tumor, Nodes, Metastasis (TNM) stage, location and the patient's general condition
8. Stage T1 and T2
9. Tumor listed N0 satisfying the following conditions (21 days validity period): A) absence of lymphadenopathy palpable on clinical examination of the ENT investigator. B) CT scan or MRI with injection of contrast product: lack of suspicious adenomegaly for metastasis = node size less than one centimeter and 1.5 cm for the group IIa, ovoid, homogeneous, not taking contrast and showing no signs of lymph perinodal invasion ( hyperdensity fat, vascular adhesion), absence of lymph node group (> 3)
10. Systematic ENT endoscopy eliminating a second synchronous tumor and precisely establishing the T (21 days validity period)
11. Absence of metastasis: M0

Exclusion criteria:

1. Failure of one of the inclusion criteria
2. Other cancer being treated
3. Non-invasive tumor: high-grade dysplasia, carcinoma in situ
4. Inadequate tumor excision: margins invaded without further recovery in safe zone
5. Contraindications to surgery such sentinel node or lymph node dissection
6. Contraindications to radiotherapy
7. Contraindications to performing a scan:

   * Known allergy or intolerance to the injected product and particularly with Technetium-99
   * Pregnancy
8. Refusal to accept the full treatment regardless of the strategy
9. Follow-up not possible
10. Refusal to accept the described follow-up and / or provide the necessary information for the study
11. Patient already treated for the tumor outside an excision biopsy
12. Patient who previously had chemotherapy or immunotherapy for another cancer outside VADS within less than 6 months
13. Patient undergoing cervical or VADS radiotherapy whatever the cause or time
14. Patient who have had cervical spine surgery regardless of the cause or time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2008-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Nodal recurrence rate | 24 months after the surgery
  The absence of recurrence at 2 years will be affirmed by the absence of clinical signs confirmed by a medical imaging exam.

SECONDARY OUTCOMES:
Evaluation of quality of life with Head and Neck 35 (H&N35) | At the inclusion, and at 2, 4, 6, 12 and 24 months after the surgery
  Evaluate quality of life on the two years of the follow up
Evaluation of the costs | At the inclusion, and at 2, 4, 6, 8, 10, 12 16, 20 and 24 months after the surgery
  The costs will be collected Under usual forms as the direct, indirect and intangible costs, directly to the relevant services and patients themselves
Evaluation of quality of life with Quality of Life Questionnaire Core 30 (QLQ-C30) | At the inclusion, and at 2, 4, 6, 12 and 24 months after the surgery
  Evaluate quality of life on the two years of the follow up
Evaluation of quality of life with EuroQOL 5D (EQ 5D) | At the inclusion, and at 2, 4, 6, 12 and 24 months after the surgery
  Evaluate quality of life on the two years of the follow up
Evaluation of quality of life with Short Form 36 (SF36)) | At the inclusion, and at 2, 4, 6, 12 and 24 months after the surgery
  Evaluate quality of life on the two years of the follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garrel R, Poissonnet G, Moya Plana A, Fakhry N, Dolivet G, Lallemant B, Sarini J, Vergez S, Guelfucci B, Choussy O, Bastit V, Richard F, Costes V, Landais P, Perriard F, Daures JP, de Verbizier D, Favier V, de Boutray M. Equivalence Randomized Trial to Compare Treatment on the Basis of Sentinel Node Biopsy Versus Neck Node Dissection in Operable T1-T2N0 Oral and Oropharyngeal Cancer. J Clin Oncol. 2020 Dec 1;38(34):4010-4018. doi: 10.1200/JCO.20.01661. Epub 2020 Oct 14. PMID 33052754